CLINICAL TRIAL: NCT01399138
Title: The Effect of Blueberry Powder Supplementation on Cardiovascular Risk Factors in Subjects With the Metabolic Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was closed on February 24, 2015.
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: U.S. Highbush Blueberry Council (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PBRC 10014
Record Dates: First submitted 2011-06-01; First posted 2011-07-21 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Metabolic Syndrome
Keywords: Pre-diabetes; Metabolic syndrome; Diabetes; Hypertension; Blueberries; Anthocyanins; Insulin sensitivity; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Diabetes Mellitus; Hypertension; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Powder (Experimental): A blueberry smoothie will be consumed at the breakfast and dinner meals.
  Interventions: Dietary Supplement: Blueberry Powder
- Placebo (Placebo Comparator): A placebo smoothie will be consumed at the breakfast and dinner meals.
  Interventions: Dietary Supplement: Blueberry Powder

INTERVENTIONS:
Dietary Supplement: Blueberry Powder — The groups will be randomized to receive 45g of blueberry powder or control (i.e., placebo) per day. Blueberry powder will be given as a smoothie to be consumed at the breakfast and dinner meals and an identical smoothie will be given as a control. The second smoothie will be consumed at least 6 hours from the first smoothie. The smoothies will be prepared in the metabolic kitchen and a week supply of frozen smoothies will be given to participants. Both the blueberry powder and control smoothie contain comparable energy and macronutrients

SUMMARY:
The purpose of this study is to examine the effects of a blueberry powder on insulin sensitivity, blood pressure, and vascular reactivity in subjects with metabolic syndrome.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States. In a large percentage of cases, the risk factors for CVD are modifiable if the responsible patient's phenotype is identified and appropriately treated. In particular, the metabolic syndrome encompasses insulin resistance, central obesity, dyslipidemia and hypertension, which are all major risk factors for CVD. These risk factors also cause underlying vascular abnormalities, i.e. endothelial dysfunction, that leads to progression of CVD. Endothelial function is the balance between vasodilating and vasoconstricting substances produced by the endothelium. Endothelial dysfunction is a common feature of insulin resistance and hypertension. In addition, endothelial dysfunction represents a very early step in the process of atherosclerosis and is associated with increased adverse CVD outcomes.

It has been well established that lifestyle modifications (changes in dietary intake and increase in physical activity) can effectively improve CVD risk factors associated with metabolic syndrome. The success of maintaining these lifestyle changes in humans over the long term is poor. Therefore, strategies to reduce prevalence of metabolic syndrome by pharmacological means have been adopted by practicing physicians. However, because of the widespread use of dietary supplements by the general public, nutritional supplementation that includes use of natural products that effectively modify the components of metabolic syndrome represent an attractive approach.

A diet rich in fruits and vegetables clearly has been shown to have significant health benefits. In particular, increased consumption of blueberries has demonstrated beneficial health effects for CVD and certain components of the metabolic syndrome, such as hypertension, insulin resistance and/or type 2 diabetes. These health benefits from blueberries may be attributable to their phenolic bioactive compounds, such as anthocyanins, which also have antioxidant properties. Although both human and animal studies demonstrated the anti-diabetic effect of blueberries, there is a paucity of data detailing the efficacy of increased blueberry consumption upon CVD risk factor modification in human subjects. Thus, given the concern regarding the ability to significantly increase and maintain an individual's fruit and vegetable consumption long-term, the role of dietary supplementation with bioactive components contained in whole blueberries becomes not only an attractive, but a feasible daily dietary intervention.

Our lab has previously shown that obese, nondiabetic and insulin-resistant human subjects that consumed blueberry powder once a day (in the form of a blueberry smoothie) for 6 weeks improved their insulin sensitivity when compared to their counterparts that consumed a placebo smoothie. Unfortunately, definitive blood pressure measurements were not conducted in this study. The investigators used a single clinic measurement which did not show any blood pressure lowering effects with consuming the blueberry smoothies. An 8-wk preclinical trialin spontaneously hypertensive stroke-prone rats, however, showed that supplementation with blueberry powder lowered systolic blood pressure. Thus, it is plausible that blood pressure lowering effects were not seen in our previous study because the investigators did not evaluate a suitable population (with hypertension) and did not use a more precise technique.

Therefore, based on the positive results in our prior human study with the use of blueberry powder increasing insulin sensitivity and given the relationship of CVD risk factors to insulin resistance, this project's overall objective is to examine the role of dietary supplementation with blueberry powder on CVD risk factors in subjects with metabolic syndrome. In particular, the investigators will evaluate changes in insulin sensitivity with the use of the frequently sampled intravenous glucose tolerance test (FSIVGTT), hypertension with the use of a precise ambulatory blood pressure monitoring system and vascular reactivity as a surrogate marker for underlying endothelial abnormalities. To our knowledge, no research studies have evaluated endothelial function and blueberries in humans. To accomplish our goal, the investigators will conduct a randomized, double-blinded and placebo-controlled clinical study with a fixed amount of blueberry powder in the form of a smoothie. The investigators hypothesize that increased daily consumption of blueberry powder will be effective in increasing insulin sensitivity, decreasing blood pressure, and improving vascular wall function in a population with metabolic syndrome that is at high-risk for CVD.

ELIGIBILITY:
Inclusion Criteria:

Men and women with metabolic syndrome and meeting all criteria listed below will be included in the study:

* Subjects ≥ 20 years of age.
* Subjects not currently treated with diabetes medication; however, Metformin use for pre-diabetes is acceptable if the subject is willing to stop taking the medication 2 weeks prior to and during the study.
* Subjects with impaired fasting glucose (100-125 mg/dL) or impaired glucose tolerance (140-199 mg/dL after 2-hr OGTT).
* Subjects with fasting insulin ≥ 10 µIU/ml.
* Subjects with a body mass index (BMI) ≥ 30 and ≤ 45.
* Subjects with hypertension: no medication (140-179 mmHg systolic or 90-109 mmHg diastolic) or currently taking antihypertensive medication.
* Written informed consent obtained PRIOR to performing any screening tests or study procedures.

Exclusion Criteria:

* Subjects with a prior history of Type 2 diabetes
* Women who are pregnant or who are lactating.
* Women of childbearing potential who are not using an effective method of birth control (i.e.,barrier method, intrauterine and cervical devices, oral contraceptives, hormonal injections (Depro Provera® ), condoms with spermicidal gel or foam, contraceptive patch (Ortho Evra), diaphragm, or abstinence), are not surgically sterilized (including tubal ligation and hysterectomy), or not at least 2 years postmenopausal. All women of childbearing potential will have a pregnancy test performed at the screening. If a subject becomes pregnant during the study, they will be dropped from the study.
* Subjects who have type 1 diabetes.
* Subjects who are currently on thiazolidinediones (rosiglitazone or pioglitazone) or who have taken these agents in the previous 12 weeks.
* Subjects who are on concomitant therapy with glucocorticoids (except topical or inhalant glucocorticoids). Other medications that have an effect on glucose homeostasis (i.e. ACE inhibitors) are acceptable if they have been administered in a stable dosage during the preceding 6 months and dosage will continue unchanged during the study.
* Subjects with a history or evidence of significant gastrointestinal dysfunction, e.g. irritable bowel syndrome; inflammatory bowel disease; ulcerative colitis or Crohn's disease; regional enteritis; diverticulosis or diverticulitis; significant gastroparesis; GI stricture, partial or complete gastrectomy or small bowel resection; autonomic neuropathy consisting of dysphasia; delayed gastric emptying or diarrhea; chronic, severe constipation; peptic ulceration, colonic ulceration, or GI bleeding.
* Subjects who have chronic use of laxatives or cathartics. The use of stool softeners is acceptable. Use of bulking agents, if required, should remain constant.
* Subjects who are taking concomitant therapy with medications known to be nephrotoxic, such as aminoglycosides, methicillin, and cyclosporin.
* Subjects who have evidence of clinically significant renal dysfunction or disease, e.g. serum creatinine >1.5 mg/dL in males and >1.4 mg/dL in females and/or BUN >50 mg/dL, proteinuria of >1 gram/day or 4+ proteinuria on dipstick urinalysis.
* Subjects with clinically significant cardiovascular dysfunction and/or history (within the preceding 6 months) of significant cardiovascular dysfunction, e.g., congestive heart failure or serious arrhythmia, myocardial infarction, cardiac surgery; transient ischemic attacks or cerebrovascular accident during the preceding six months; diagnosis of symptomatic autonomic neuropathy with a history of orthostatic hypertension, syncope, or hypertension with a systolic blood pressure of ≥180 mm Hg or diastolic blood pressure ≥110 mm Hg at the time of screening visit.
* Subjects who have evidence within the preceding 6 months of hepatic disease or dysfunction, e.g. AST, ALT, alkaline phosphatase or total bilirubin twice the upper limit of normal; hepatitis; jaundice; cirrhosis.
* Subjects with clinically significant pulmonary, neurologic, hematologic, immunologic, neoplastic or metabolic disease.
* Subjects with evidence or recurrence of malignancy within the past five years, other than excised basal cell carcinoma.
* Subjects for whom surgery is anticipated during the study period.
* Subjects with a history of substance abuse or alcoholism within the past 5 years, or significant psychiatric disorder that would interfere with the subject's ability to complete the study.
* Subjects who have donated blood during the month prior to study entry or planned during the study.
* Subjects who have participated in other studies using an investigational drug during the preceding 3 months.
* Subjects who are current smokers or have smoked within the previous 6 months. No smoking will be allowed during the study.
* Subjects who are allergic to blueberries.
* Subjects who are allergic to red dye or blue dye food coloring.
* Subjects who are lactose intolerant.
* Subjects who consume and drink daily servings of berries (i.e., blueberries, strawberries, bilberries, cranberries, elderberries, and raspberries), grapes, fruit juices that contain berries and grapes, and wine more than 3 times per week.
* Subjects that have had a fluctuation in body weight >5% in the preceding 2 months.
* Subjects who are taking prescription or over the counter medication or supplements for desired weight loss.
* Subjects that have peripheral vascular disease in the arms.
* Subjects that have a history of blood clots.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Systolic and Diastolic Blood Pressure at 6 weeks | Baseline and Week 6 (The study has 6 weeks)
  This procedure records your blood pressure and heart rate. You will wear a device the size of a small camera connected to a blood pressure cuff on your arm for a period of seven days. The cuff of this device inflates automatically every 30 minutes during the day and every 60 minutes during the night. Upon inflation, the device will make a quiet noise and will cause pressure on your arm. At the end of the seven days, you will return to the clinic or Inpatient Unit at Pennington to have the monitor removed. Depending upon the amount of data collected, you may be asked to wear the monitor for additional days.

SECONDARY OUTCOMES:
Change from Baseline in Response of Blood Vessels to a Stimulus at 5 weeks | About 1 hour (Baseline and at Week 5)
  This procedure is performed to determine the response of your blood vessels to a stimulus. You will lie on your back on a bed and have a blood pressure cuff placed on your non-dominant arm (the arm you do not write with). Probes will be attached to the index finger on both of your hands, and these probes will be slightly inflated to be held in place. The blood pressure cuff will be inflated for five minutes. It will then be deflated rapidly. Data will be recorded continuously throughout the test. The entire procedure will take approximately 1 hour.
Change from Baseline in insulin sensitivity at 6 weeks | About 5 hours(Baseline and Week 6)
  This test measures how well your body produces insulin in response to a sugar challenge. Insulin is normally produced in your body during meals and helps your body use sugar. There will be 2 IV lines, one line inserted into a vein in each of your arms. After collecting a baseline sample of your blood we will inject a solution containing sugar into one of the IV lines. We will then monitor your blood sugar and insulin levels by drawing blood from the other IV for 20 minutes. After 20 minutes we will inject insulin into the IV line and we will continue to monitor your blood sugar and insulin levels for another 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: William T Cefalu, MD, Principal Investigator — Pennington Biomedical Research Center; April J Stull, Ph.D., Study Director — Pennington Biomedical Researcher
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States